CLINICAL TRIAL: NCT04715568
Title: Occult Cardiovascular Disease With Chronic Exposure to Secondhand Tobacco Smoke
Brief Title: Secondhand Tobacco Smoke and Cardiovascular Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-30189
Record Dates: First submitted 2020-12-17; First posted 2021-01-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: Second Hand Tobacco Smoke
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Losartan; Angiotensin Receptor Antagonists; Antihypertensive Agents

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled crossover clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, research staff, and subjects, with the exception of the San Francisco Veteran's Administration (VA) Medical Center Research Pharmacist, will be blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo then Losartan (Experimental): Placebo tablets will be administered for the first 4 weeks followed by a washout period of 2 weeks. After the washout period has been completed, losartan tablets will be administered for the next 4 weeks.
  Interventions: Drug: Losartan; Drug: Placebo
- Losartan then Placebo (Experimental): Losartan tablets will be administered for the first 4 weeks followed by a washout period of 2 weeks. After the washout period has been completed, placebo tablets will be administered for the next 4 weeks.
  Interventions: Drug: Losartan; Drug: Placebo

INTERVENTIONS:
Drug: Losartan — 50 mg tablets taken orally
  Other Names: Cozaar; Angiotensin II Receptor Blocker; Antihypertensive
Drug: Placebo — Tablets taken orally
  Other Names: Inactive drug

SUMMARY:
This is a double-blind randomized placebo-controlled crossover clinical trial of efficacy and safety of an FDA-approved angiotensin receptor blocker (losartan) to improve cardiopulmonary outcomes in individuals with pre-Chronic Obstructive Pulmonary Disease (COPD) due to prolonged exposure to secondhand tobacco smoke.

DETAILED DESCRIPTION:
Secondhand tobacco smoke (SHS) remains a major public health problem.This is important particularly as the generations that endured the highest amount of SHS exposure are aging, which could potentially accentuate the SHS-related occult health problems that may have been previously too subtle to be recognized. Although acute and subacute health effects of exposure to SHS have been studied, its long-term consequences have been more difficult to examine in part due to challenges with exposure assessment. Nonsmoking flight attendants (FA) who worked on commercial aircrafts before the enactment of the smoking ban were exposed to heavy SHS in aircraft cabin for many years, in a range similar to the nicotine exposure burden experienced by "light" smokers. The regularity of this intense exposure in the cabin work environment lends itself to relatively accurate SHS exposure quantification through employment history, and makes the exposed FA a unique population in which the long-term health effects of previous exposure to SHS could be examined as a form of "natural" experiment that is also generalizable to other SHS exposed populations.

Over the past several years, the investigators recruited a nonsmoking cohort of FA with such history of cabin SHS exposure who had subclinical signs and symptoms of pulmonary disease. Furthermore, while the FA in this cohort had no history of known cardiovascular disease, and were able to perform well on maximum effort exercise testing, they had an abnormal cardiovascular (hypertensive) response to exercise (HRE) that was associated with their cabin SHS exposure. Subtle abnormal cardiovascular response to exercise in the absence of overt disease, such as what the investigators observed in this cohort, has been described in other populations with likely subclinical disease and is suggested to be associated with impaired cardiovascular function with potential future adverse outcomes. However, the underlying mechanisms that contribute to these abnormal cardiovascular responses are unclear, and the rationale for initiation of preventative medical interventions in this setting remains unproven. Thus, the nature and clinical significance of these subtle abnormalities demands further investigation.

The hypothesis of this study is that:

1. Prolonged exposure to secondhand tobacco smoke (SHS), even when remote, is associated with occult cardiovascular disease as determined by (a) abnormal cardiac structure and function, (b) abnormal vascular structure and function, and (c) abnormal circulatory mediators, which altogether generate a hypertensive response to exertion and limit exercise capacity.
2. Management of hypertensive response to exercise (HRE) via blocking of the renin-angiotensin system, using an angiotensin-converting enzyme (ACE) receptor blocker, reduces the hypertensive response and improves exercise capacity, proxies for long-term cardiovascular health outcomes.

The investigators will investigate the above hypothesis through the following specific aims:

Specific Aim 1- Determine whether hypertensive response to exercise (HRE) is associated with abnormal cardiac and/or vascular structure and function in flight attendants (FA) with prolonged cabin SHS exposure but without overt cardiovascular disease. The investigators will perform cardiac magnetic resonance imaging (MRI) to measure myocardial dimensions and function including left ventricular (LV) mass, volume, ejection fraction (LVEF), and diastolic function. The investigators will also measure aortic stiffness by regional pulse wave velocity (PWV) measurement in the thoracic aorta from the MRI. The investigators will then examine the associations of these outcomes with SHS exposure and HRE.

Specific Aim 2- Determine whether HRE is associated with abnormal circulatory markers of cardiovascular disease in those with prolonged SHS exposure but without overt disease. The investigators will examine subjects' peripheral blood samples for circulatory markers of systemic inflammation, vascular function, and prothrombotic state including ACE, C-reactive protein (CRP), endothelin-1 (ET-1), P-selectin, fibrinogen, and von Willebrand Factor (vWF). Moreover, the investigators will perform molecular phenotyping of peripheral blood monocytes, an important culprit in atherogenesis, using mass cytometry in search for a proinflammatory profile associated with cardiovascular disease. The investigators will then examine the associations of these outcomes with HRE and SHS exposure.

Specific Aim 3- Determine whether short-term treatment with an ACE receptor blocker (Losartan) improves HRE and exercise capacity in those with prolonged exposure to SHS but without overt cardiovascular disease. The investigators will perform a placebocontrolled double-blind randomized controlled trial (RCT) in subjects with HRE but without known cardiovascular disease to determine the efficacy (and safety) of blocking the reninangiotensin system in reducing HRE and improving exercise capacity, a proxy for improved cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and provide informed consent.
* Adults >= 40 years of age.
* Must have a history of occupational exposure to secondhand tobacco smoke for at least 5 years such as flight attendants who worked for airlines before the smoking ban on aircrafts went into effect or casino workers who worked at casinos with no smoke-free policies.
* Must have never smoked or have a remote history of light smoking defined as follows:

  * Lifetime smoking history equivalent to < 1 pack-year and
  * No smoking history for >= 20 years at the time of enrollment.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* Subject is pregnant, breast-feeding, or plans to become pregnant.
* Current therapy with angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB).
* Known intolerance to ACE inhibitor or ARB.
* History of angioedema.
* Conventional indication for ACE inhibitor or ARB (e.g., history of myocardial infarction, known cardiomyopathy).
* Blood pressure less than 90 mm Hg systolic or 60 mm Hg diastolic while standing or sitting.
* Known unilateral or bilateral renal artery stenosis higher than 70%.
* Renal insufficiency (Creatinine Clearance <30 mL/min by Cockcroft-Gault calculation).
* Current regular use of NSAIDs defined as daily use on 5 or more days of the week for more than one month.
* Potassium supplementation or serum potassium level of 5.0 milliequivalents (mEq)/dL or higher at V1.
* Current use of a potassium sparing diuretic.
* History of clinically overt cardiovascular disease including: stable or unstable angina; chest discomfort and dyspnea with baseline exertion; symptomatic coronary artery disease (as defined by history of abnormal stress test; cardiac catheterization showing >70% coronary artery stenosis; history of revascularization; pathologic Q waves on EKG); poorly controlled resting hypertension (SBP>160/ DBP>95); congestive heart failure (CHF) (as defined by left ventricular ejection fraction (LVEF) <55%; physical exam findings of CHF; symptomatic pulmonary edema); significant (>mild) valvular heart disease; congenital heart disease; cardiac arrhythmias including frequent premature atrial or ventricular contractions (>5 per minute).
* History of clinically overt pulmonary disease that may interfere with study procedures, including: greater than mild asthma, COPD, emphysema, chronic interstitial lung disease, and pulmonary hypertension.
* Neuromuscular disorders or physical disability to perform exercise testing using an ergometer.
* Significant history of recreational drug use other than marijuana as defined by: recreational drug use within the last 30 years of recruitment (or) recreational drug use at a frequency of more than once a month before 30 years.
* Marijuana use more than once a week.
* Other uncontrolled chronic illnesses which in the judgment of the study physician would interfere with completing study procedures.
* Failure to keep screening appointments or other indicators of non-adherence.
* Concomitant participation in another interventional study.
* Subjects with BMI <15 or >40 kg/m2.
* MRI Scan Participation Exclusion Criteria - The participants will be excluded from the MRI portion of the study if they have a metallic object embedded or implanted in their body that is incompatible with Magnetic Resonance (MR) scanning, including MR incompatible pacemaker or defibrillator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Left Ventricular Ejection Fraction (LVEF) | Baseline, approximately 1 day
  LVEF will be measured using Magnetic Resonance Imaging (MRI) using General Electric 1.5 Tesla MRI system without gadolinium contrast. In accordance with the American College of Cardiology (ACC), results will be reported quantitatively and qualitatively as follows: Hyperdynamic = LVEF greater than 70%, Normal = LVEF 50% to 70% (midpoint 60%), Mild dysfunction = LVEF 40% to 49% (midpoint 45%), Moderate dysfunction = LVEF 30% to 39% (midpoint 35%), Severe dysfunction = LVEF less than 30%.
Mean Aortic pulse wave velocity (PWV) | Baseline, approximately 1 day
  Aortic pulse wave velocity (PWV) is a marker of aortic stiffness and will be measured (in meters/second) by regional PWV measurement in the thoracic aorta from the MRI (General Electric 1.5 Tesla MRI system without gadolinium contrast).
Change in Prevalence of CD14++CD16- | Up to 10 weeks
  CD14++CD16- are markers of pro-inflammatory phenotypes that will be measured among peripheral blood monocytes using mass cytometry.
Change in Mean Peak Oxygen Consumption (VO2 Peak) Level | Up to 10 weeks
  VO2 Peak is the peak rate of oxygen consumption in milliliters per kilogram per minute (mL/(kg·min) measured during incremental exercise on a Cardio-Pulmonary Exercise Test (CPET). Patients are encouraged to exercise to their maximum endurance or until the nurse ends exercise due to symptoms like pain, dizziness, syncope, excessive dyspnea, or leg discomfort.

SECONDARY OUTCOMES:
Mean Left Ventricular Mass | Baseline, approximately 1 day
  Left ventricular mass will be measured (in grams/m2) using cardiac MRI (General Electric 1.5 Tesla MRI system without gadolinium contrast).
Mean Left Ventricular Volume | Baseline, approximately 1 day
  Left ventricular volume will be measured (in mL) using cardiac MRI (General Electric 1.5 Tesla MRI system without gadolinium contrast).
Change in Mean Angiotensin Converting Enzyme (ACE) Level | Up to 10 weeks
  ACE is a central component of the renin-angiotensin system (RAS), which controls blood pressure by regulating the volume of fluids in the body. Level of ACE will be measured in micrograms per liter from peripheral blood sample.
Change in Mean C-Reactive Protein (CRP) Level | At baseline assessment (V1); 4th week of V2 (placebo/losartan) treatment period; and 4th week of V3 (placebo/losartan) treatment period
  CRP is an acute phase reactant and will be measured (in mg/L) from peripheral blood sample.
Change in Mean Endothelin-1 Level | Up to 10 weeks
  Endothelin-1 is a potent vasoconstrictor produced by vascular endothelial cells and will be measured from peripheral blood sample.
Change in Mean P-selectin Level | Up to 10 weeks
  P-selectin is a transmembrane glycoprotein that functions as a cell adhesion molecule on the surfaces of activated endothelial cells and will be measured from peripheral blood sample.
Change in Mean Fibrinogen Level | Up to 10 weeks
  Fibrinogen is a glycoprotein that plays a pivotal role in normal homeostasis as a substrate for conversion to fibrin and a facilitator of wound healing. It will be measured in milligrams per deciliter from peripheral blood sample.
Change in Mean von Willebrand Factor (VWF) | Up to 10 weeks
  VWF is a large multimeric glycoprotein that performs critical functions in primary hemostasis. It will be measured in micrograms per deciliter from peripheral blood sample.
Change in Mean Maximum Workload | Up to 10 weeks
  The maximum amount of workload achieved (in watts) during an incremental CPET.
Change in Mean Maximum Oxygen Pulse | Up to 10 weeks
  Oxygen pulse is the ratio between Oxygen consumption (VO2) and heart rate. The maximum O2-pulse (mL/beat), a proxy for stroke volume, will be measured during incremental CPET.
Change in Mean Slope of Systolic Blood Pressure (SBP) | Up to 10 weeks
  The rate at which the SBP increases over the workload achieved in watts during an incremental CPET is the Slope of SBP.
Change in Mean Slope of Diastolic Blood Pressure (DBP) | Up to 10 weeks
  The rate at which the DBP increases over the workload achieved in watts during an incremental CPET is the Slope of DBP.
Change in Mean Slope of Heart Rate (HR) | Up to 10 weeks
  The rate at which the HR increases over the workload achieved in watts during an incremental CPET is the Slope of HR.
Change in Mean Change in Borg Score | Up to 10 weeks
  Borg Rating of perceived exertion is a widely used and reliable indicator to monitor and guide exercise intensity. The scale allows individuals to subjectively rate their level of exertion during exercise testing. The revised category-ratio scale (0 to 10 scale) will be used, where 0 indicates no perceived exertion and 10 indicates maximal perceived exertion.
Change in Mean Moderate-to-Vigorous Physical Activity (MVPA) | Up to 10 weeks
  MVPA is measured with Metabolic Equivalents (METs). A MET is the ratio of a person's working metabolic rate compared to their resting metabolic rate. MVPA is any activity over 3 METs. An Actigraph monitor will be used to measure MVPA.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Arjomandi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans' Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of California, San Francisco (UCSF) website for Arjomandi Lab — https://arjomandilab.ucsf.edu/